CLINICAL TRIAL: NCT01014455
Title: Monitoring of Exhaled Carbon Monoxide to Promote Pre-operative Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: David O. Warner, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-006998
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Results first posted 2011-08-22 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-07

CONDITIONS: Smoking
Keywords: surgery
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CO reminder (Experimental): A brief intervention that recommends preoperative fasting from cigarettes and that informs patients that their smoking status will be checked before surgery using inhaled CO monitoring will decrease their exposure to cigarette smoke prior to surgery
  Interventions: Behavioral: Informing surgical patients about CO monitoring
- no CO reminder (Placebo Comparator): a brief intervention that recommends fasting but does not mention that CO will be checked
  Interventions: Behavioral: a brief intervention recommending preoperative abstinence from smoking

INTERVENTIONS:
Behavioral: Informing surgical patients about CO monitoring — A brief intervention that recommends preoperative fasting from cigarettes and that informs patients that their smoking status will be checked before surgery using inhaled CO monitoring will decrease their exposure to cigarette smoke prior to surgery
  Arms: CO reminder
Behavioral: a brief intervention recommending preoperative abstinence from smoking — a brief intervention that recommends fasting but does not mention that CO will be checked
  Arms: no CO reminder

SUMMARY:
Smoking causes 90% of all lung cancer deaths among men and 80% of lung cancer deaths in women. Surgery is a great opportunity to help patients quit smoking. Smokers are at increased risk for heart, lung, and wound complications around the time of surgery. Even a brief abstinence from smoking can produce benefits. Surgery can also motivate smokers to quit spontaneously. If the investigators can take advantage of this great opportunity, they may be able to help many smokers quit using simple means. However, currently most smokers continue to smoke cigarette on the morning before surgery, as shown by the measurement of exhaled carbon monoxide (CO) on the morning of surgery. CO is one of the many poisons in cigarette smoke. It only stays in the body for a few hours. By asking smokers to blow into a small machine, the investigators can test the CO level in the smokers' body and thus know if they have just smoked within the past few hours. The goal of this study is to determine the role of carbon monoxide monitoring as a means to decrease cigarette smoking before surgery. The investigators will identify a group of smokers who are scheduled for surgery and invite them to participate. One or two days before surgery, half of the patients will receive a brief advice about quit smoking. The other half of patients will be told that their CO will be checked before surgery, in addition to the brief advice. On the morning of surgery, the investigators will then check their CO level to determine if they have followed the advice. In order to have a better understanding about the factors influencing patients' intent to quit smoking, the investigators will ask all study participants to fill out a questionnaire. The questionnaire is constructed according to behavioral theories which provide good framework for studying people's intent and behavior. If the investigators are successful, they will determine how much of an impact the message of CO testing has on smoking before surgery. The investigators will also gain insights into facilitators and barriers to smoking cessation around the time of surgery. The brief intervention evaluated in this study has potential to be disseminated and to promote the long term health of surgical patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 yrs. scheduled for elective non-cardiac surgery at Mayo Clinic Rochester;
2. Current smoking, defined as > 100 cigarettes lifetime consumption and self-report of smoking every day.

Exclusion Criteria:

1. An inability to understand consent procedures;
2. Inability to complete a written questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Warner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Shi Y, Ehlers S, Warner DO. The theory of planned behavior as applied to preoperative smoking abstinence. PLoS One. 2014 Jul 24;9(7):e103064. doi: 10.1371/journal.pone.0103064. eCollection 2014. PMID 25057969
- [Derived] Shi Y, Ehlers S, Hinds R, Baumgartner A, Warner DO. Monitoring of exhaled carbon monoxide to promote preoperative smoking abstinence. Health Psychol. 2013 Jun;32(6):714-7. doi: 10.1037/a0029504. Epub 2012 Aug 27. PMID 22924451

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cigarette smokers scheduled for elective non-cardiac surgery were recruited from the preoperative evaluation clinic at Mayo Clinic Rochester.
Pre-assignment Details: Inform consent was obtained after data collection(approved by the IRB) because informing patients of the study at time of enrollment would have required providing information making it impossible to evaluate the hypothesis. Study records from patients who declined informed consent (n=14) were destroyed and are not included in the analysis.
Period: Overall Study
Arm/Group | CO Reminder | no CO Reminder
Started | 82 | 87
Completed | 82 | 87
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CO Reminder | no CO Reminder | Total
Number analyzed (Participants) | 82 | 87 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 70 | 136
  >=65 years | 16 | 17 | 33
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (12) | 53 (12) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 47 | 87
  Male | 42 | 40 | 82
Region of Enrollment [Number; unit: participants]
  United States | 82 | 87 | 169

OUTCOME MEASURES:

1. Primary Outcome: Preoperative Carbon Monoxide Levels
Time Frame: the morning of surgery
Reporting Status: Not Posted

2. Primary Outcome: Exhaled CO Level Measured Immediately Prior to Surgery
Description: On the morning of surgery, as matter of clinical routine all patients receiving surgery requiring anesthesia services at one of the two main surgical facilities at Mayo Clinic Rochester and who self-report as a current smoker are asked about their typical cigarette consumption (cigarettes per day), if they have smoked cigarettes today, and have their exhaled CO levels measured (Micro Smokerlyzer; Bedfont, United Kingdom). This information is entered into the clinical record. The CO monitors are maintained by the Division of Respiratory Therapy, including regular calibration.
Time Frame: The median time from study assessment at POE to surgery was 1 day with an interquartile range of 1 to 3 days.
Population: 5 participants did not complete CO measures and were excluded from the analysis of primary outcome
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | CO Reminder | no CO Reminder
Number analyzed (Participants) | 80 | 84
ppm | 9.7 (8.0) | 9.3 (6.6)
Statistical Analysis 1: Comparison: CO Reminder vs no CO Reminder; Test type: Superiority or Other; p = 0.672, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | CO Reminder | no CO Reminder
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study subjects received the additional questionnaire on smoking behavior, which itself could heighten awareness of perioperative tobacco use issues and could be viewed as an additional intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes